CLINICAL TRIAL: NCT06904638
Title: Underprescribing in Geriatric Patients: a Prevalence Study and Analysis of Factors Contributing to Potential Prescription Omissions (Under-PRES)
Acronym: Under-PRES
Status: Recruiting | Type: Observational
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Other Study IDs: INRCA_004_2025
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Older People
Keywords: underprescription; START criteria; potential prescriptive omissions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- older adults: Geriatric patients admitted to a geriatric hospital unit or attending an outpatient geriatric clinic

SUMMARY:
This observational study will determine the prevalence of underprescription in a cohort of elderly patients, recruited at the time of an outpatient geriatric visit, or hospitalized, upon admission to a geriatric ward.

DETAILED DESCRIPTION:
Polypharmacy in older patients is associated with both inappropriate drug prescribing and underprescription or omission of appropriate medications. Potential prescriptive omission (PPO), defined as the underprescription of potentially beneficial drugs, is increasing across all care settings and is associated with adverse clinical outcomes. However, in some cases, PPO may represent a legitimate medical decision.

The aim of this study is to investigate the phenomenon of underprescription by differentiating between justified and inappropriate potential prescriptive omissions (PPOs) in elderly patients in both hospital and outpatient settings, using the Screening Tool to Alert to Right Treatment (START) criteria, version 3.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric ward admission or outpatient geriatric appointment
* Capacity to provide informed consent by the patient or legal guardian

Exclusion Criteria:

* Limited life expectancy as measured by the Clinical Frailty Scale (CFS) >8

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients at admission to a geriatric ward or at the time of outpatient geriatric visits
Sampling Method: Non-Probability Sample
Enrollment: 374 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of potential prescription omissions (PPOs) | at baseline and 3 months later
  Prevalence of potential prescription omissions (PPOs) will be evaluated by Screening Tool to Alert doctors to Right Treatment (START) criteria version 3 in aged patients enrolled on admission to geriatric departments of participating centers or during geriatric outpatient clinic visits

SECONDARY OUTCOMES:
Characterisation of the potential prescription omissions (PPOs) | at baseline and 3 months later
  The reasons for underprescription will be investigated to differentiate between justified and inappropriate potential prescriptive omissions (PPOs). Patients and/or their family members and/or the general practitioner will be interviewed to assess the potential reasons related to underprescription.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cherubini, MD, Study Chair — IRCCS INRCA, Ancona, Italy
Locations (2):
- Italy (2):
  - IRCCS INRCA Hospital, Ancona
  - IRCCS INRCA Hospital, Cosenza

IPD SHARING:
Plan to Share IPD: No